CLINICAL TRIAL: NCT04352842
Title: Cardiac Structural and Functional Characteristics in COVID-19: A Dynamic Echocardiographic Study
Brief Title: Echocardiographic Manifestation in Patient With COVID-19 （EARLY-MYO COVID-19）
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COVID19-Echocardiography
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-04

CONDITIONS: Covid19; Echocardiography
Keywords: COVID-19; Echocardiography; cardiac structure; cardiac function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-survivors: Patients deceased during the study period
  Interventions: Other: Echocardiography
- Survivors: Patients survived during the study period
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — An expert with 17-year professional experience performed all the echocardiography examinations using a GE LOGIQTM e portable color ultrasound diagnostic machine (GE Healthcare, WI, USA) that was specially used in the contaminated area. Two-dimensional and Doppler echocardiographic measurements were conducted following the recommendations of the American Society of Echocardiography

SUMMARY:
The cardiovascular effects of coronavirus disease 2019 (COVID-19) are not yet fully known. We conducted a prospective and dynamic echocardiographic study to investigate the cardiac structural and functional changes in COVID-19 patients in intensive care unit (ICU).

DETAILED DESCRIPTION:
The ongoing pandemic of coronavirus disease 2019 (COVID-19) caused by the newly discovered severe acute respiratory syndrome coronavirus 2 (SAR-CoV-2) has become a global health crisis, resulting in 3,435,894 confirmed infections and 239,604 deaths worldwide by 4 May 2020 1. Although acute respiratory syndrome is the main manifestation of the disease2, the understanding of the impact of the virus on other organs is of importance in terms of multiple organ dysfunction/failure that contributed to the increased mortality in patients with COVID-19.

With the increase of confirmed cases and the accumulation of clinical data, the cardiovascular manifestations caused by COVID-19 has raised concern3. Some studies have reported that a certain percentage of patients presented cardiac injury as indicated by elevated cardiac biomarkers such as high-sensitivity cardiac troponin-I (hs-cTnI) and brain natriuretic peptide (BNP) 2,4,5. Cardiac complications, including acute heart failure, cardiac rupture and even sudden cardiac arrest, has also been described in several case reports 6-8. However, autopsy studies failed to find the evidence of direct assaults by the virus in myocyte or apparent myocyte necrosis/apoptosis in the heart 9. Typical pathological finding reported was mononuclear inflammatory infiltration in the myocardial interstitium but no substantial damage in cardiomyocytes in the heart 10,11. Thus, a significant gap exists in our knowledge between the clinical investigation and postmortem findings. At present, the in vivo morphological and functional features of cardiac injury remain unknown.

We therefore performed a prospective and dynamic echocardiography study to investigate the cardiac structural and functional changes in patients with COVID-19 who were admitted to intensive care unit (ICU), and to compare the cardiac characteristics between deceased and survived patients.

ELIGIBILITY:
Inclusion Criteria:

Patients had been diagnosed of COVID-19 according to the criteria established by the WHO interim guidance and admitted to ICU because of severe or critical condition

Exclusion Criteria:

Patients who were < 18 years and whose entire stay in hospital lasted for < 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in an intensive care unit (ICU) during February 22 to April 3, 2019 in a special hospital for COVID-19 patients in Wuhan, China
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Death | From admission to April 8 2020 (cutoff day)
  Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, M.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China